CLINICAL TRIAL: NCT01862887
Title: A Phase 1, Randomized, Placebo-And Positive-Controlled Crossover Study To Determine The Effect Of A Single-Dose Of PH-797804 On QTc Interval In Healthy Volunteers
Brief Title: A Study to Investigate the Effect of PH-797804 on QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A6631035
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
MeSH Terms: interventions — PH 797804; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PH-797804 (Experimental): Subjects will receive a single 24 mg dose in the fed state
  Interventions: Drug: PH-797804
- Moxifloxacin (Experimental): Subjects will receive a single 400 mg dose in the fed state
  Interventions: Drug: Moxifloxacin
- Placebo (Experimental): Subjects will receive a single placebo dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH-797804 — Tablet, 24 mg, single dose
  Arms: PH-797804
Drug: Moxifloxacin — Tablet, 400 mg, single dose
  Arms: Moxifloxacin
Drug: Placebo — Tablet, PH-797804 matched placebo, single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of PH-797804 following dosing of a 24 mg oral tablet on the QTc interval

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy female subjects of non-child bearing potential between the ages of 18 and 55 years (inclusive). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for males.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
QTcF Interval | -1.5,-1,-0.5,0.5,2,4,5,6,7,8,12,24 hours post-dose
  QT interval corrected for heart rate using Fredericias correction

SECONDARY OUTCOMES:
QTcI Interval | -1.5,-1,-0.5,0.5,2,4,5,6,7,8,12,24 hours post-dose
  QT interval using individual heart rate correction
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 0,0.5,2,4,5,6,7,8,12,24 hours post-dose
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Maximum Observed Plasma Concentration (Cmax) | 0,0.5,2,4,5,6,7,8,12,24 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,0.5,2,4,5,6,7,8,12,24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631035&StudyName=A%20Study%20to%20Investigate%20the%20Effect%20of%20PH-797804%20on%20QTc%20Interval